CLINICAL TRIAL: NCT03760198
Title: A Phase III, Randomized, Double-Blind, Placebo Controlled, Multi-Center Study to Evaluate the Efficacy and Safety of MEDITOXIN in Treatment of Primary Axillary Hyperhidrosis
Brief Title: Evaluate the Efficacy and Safety of MEDITOXIN in Treatment of Primary Axillary Hyperhidrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT01-KR17PAH311
Record Dates: First submitted 2018-11-29; First posted 2018-11-30 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Hyperhidrosis Primary Focal Axilla
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- botulinum toxin type A (Experimental)
  Interventions: Drug: Meditoxin
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Meditoxin — 50U of MEDITOXIN is injected intradermally to each axilla
  Arms: botulinum toxin type A
Other: Placebo — normal saline is injected intradermally to each axilla
  Arms: Placebo

SUMMARY:
This study is intented to evaluate the efficacy and safety of MEDITOXIN compared to placebo in treatment of primary axillary hyperhidrosis.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged from 20 to 65, with persistent bilateral primary axillary hyperhidrosis

Exclusion Criteria:

* those who have secondary hyperhidrosis
* those who have systemic neuromuscular junction disorders
* women who are pregnant or lactating

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
the proportion of treatment responder | 4 weeks after the injection
  subjects who reported at least a 2-point improvement from baseline HDSS score

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University St. Paul Hospital, Seoul, Dongdaemun-gu, South Korea